CLINICAL TRIAL: NCT00626392
Title: Multicenter, Randomized, Double-Blind, Parallel, Acetylsalicylic Acid (ASA) Run-In Study to Evaluate the EFFECTS of Acetylsalicylic Acid on Niaspan®-Induced Flushing in Subjects With Dyslipidemia
Brief Title: Study to Evaluate the EFFECTS of Acetylsalicylic Acid (ASA) on Niaspan®-Induced Flushing in Subjects With Dyslipidemia
Acronym: ASA EFFECTS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Scott Krause, Associate Director, Abbott
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M10-241
Record Dates: First submitted 2008-02-21; First posted 2008-02-29 (Estimated); Results first posted 2009-08-25 (Estimated); Last update posted 2009-09-02 (Estimated); Status verified 2009-08

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — Niacin; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- NER 500; ASA run-in, ASA coadmin (Experimental): Aspirin (ASA) daily during run-in (1 week); ASA 30 min prior to niacin extended-release ([NER], 500 mg starting dose), daily during coadministration period (4 weeks)
  Interventions: Drug: niacin extended-release (NER); Drug: aspirin (ASA)
- NER 500; ASA Pbo run-in, ASA coadmin (Experimental): Aspirin placebo (ASA Pbo) daily during run-in (1 week); ASA 30 min prior to niacin extended-release ([NER], 500 mg starting dose), daily during coadministration period (4 weeks)
  Interventions: Drug: niacin extended-release (NER); Drug: aspirin (ASA); Drug: aspirin placebo (ASA Pbo)
- NER 500; ASA Pbo run-in, ASA Pbo coadmin (Experimental): Aspirin placebo (ASA Pbo) daily during run-in (1 week); ASA Pbo 30 min prior to niacin extended-release ([NER], 500 mg starting dose), daily during coadministration period (4 weeks)
  Interventions: Drug: niacin extended-release (NER); Drug: aspirin placebo (ASA Pbo)
- NER 1000; ASA run-in, ASA coadmin (Experimental): Aspirin (ASA) daily during run-in (1 week); ASA 30 min prior to niacin extended-release ([NER], 1000 mg starting dose), daily during coadministration period (4 weeks)
  Interventions: Drug: niacin extended-release (NER); Drug: aspirin (ASA)
- NER 1000; ASA Pbo run-in, ASA coadmin (Experimental): Aspirin placebo (ASA Pbo) daily during run-in (1 week); ASA 30 min prior to niacin extended-release ([NER], 1000 mg starting dose), daily during coadministration period (4 weeks)
  Interventions: Drug: niacin extended-release (NER); Drug: aspirin (ASA); Drug: aspirin placebo (ASA Pbo)
- NER 1000; ASA Pbo run-in, ASA Pbo coadmin (Experimental): Aspirin placebo (ASA Pbo) daily during run-in (1 week); ASA Pbo 30 min prior to niacin extended-release ([NER], 1000 mg starting dose), daily during coadministration period (4 weeks)
  Interventions: Drug: niacin extended-release (NER); Drug: aspirin placebo (ASA Pbo)

INTERVENTIONS:
Drug: niacin extended-release (NER) — Tablets administered once daily; titrated to 2000 mg maximum dose during coadministration period
  Other Names: Niaspan
Drug: aspirin (ASA) — 325 mg tablets administered once daily
  Other Names: acetylsalicylic acid
  Arms: NER 1000; ASA Pbo run-in, ASA coadmin; NER 1000; ASA run-in, ASA coadmin; NER 500; ASA Pbo run-in, ASA coadmin; NER 500; ASA run-in, ASA coadmin
Drug: aspirin placebo (ASA Pbo) — Tablets administered once daily
  Other Names: placebo
  Arms: NER 1000; ASA Pbo run-in, ASA Pbo coadmin; NER 1000; ASA Pbo run-in, ASA coadmin; NER 500; ASA Pbo run-in, ASA Pbo coadmin; NER 500; ASA Pbo run-in, ASA coadmin

SUMMARY:
The primary purpose of this study was to assess the effect of aspirin (ASA) on niacin extended-release (NER)-induced flushing in subjects with dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18 years of age or older.
* If female, subject is either not of childbearing potential, defined as postmenopausal for at least one year or surgically sterile, or is of childbearing potential and must agree to practice birth control for the duration of the study.
* Have dyslipidemia as demonstrated by laboratory results.

Exclusion Criteria:

* Have glycosylated hemoglobin (HbA1c) >/= 9.0%.
* Have nephrotic syndrome, dysproteinemias, or severe renal failure (glomerular filtration rate [GFR] < 30 mL/minute, as calculated from creatinine clearance).
* Have had unstable angina or an acute myocardial infarction (MI) within three months of the Screening Visit.
* Have had severe peripheral artery disease as evidenced by intermittent claudication within three months of the Screening Visit.
* Have had uncontrolled cardiac arrhythmias within three months of the Screening Visit.
* Have symptomatic heart failure defined as dyspnea at rest or with exertion (mild peripheral edema is not exclusionary).
* Have a systolic blood pressure measurement of > 180 mmHg or a diastolic blood pressure measurement of > 110 mmHg at the Screening or Baseline Visit.
* Have active gout or uric acid >/= 11 mg/dL.
* Have a history of hepatitis (acute or chronic), obstructive liver disease, or alanine aminotransferase (ALT; serum glutamic pyruvic transaminase [SGPT]) or aspartate aminotransferase (AST; serum glutamic oxaloacetic transaminase [SGOT]) values >/= 1.3 times the upper limit of normal (ULN) at the Screening Visit.
* Have creatine phosphokinase (CPK) >/= 3 x ULN at the Screening Visit.
* Have used an investigational study drug or participated in an investigational study within 30 days of the Screening Visit.
* Have a health condition or laboratory abnormality (inclusive of clinically significant laboratory results at Screening Visit), which, in the opinion of the Investigator, may be adversely affected by the procedures or study medications in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2008-02; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roopal Thakkar, MD, Study Director — Abbott
Locations (25):
- United States (25):
  - Huntsville, Alabama
  - Scottsdale, Arizona
  - Tucson, Arizona
  - Anaheim, California
  - Los Angeles, California
  - Newport Beach, California
  - Stockton, California
  - Vista, California
  - Westlake Village, California
  - Coral Gables, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Pembroke Pines, Florida
  - West Palm Beach, Florida
  - North Dartmouth, Massachusetts
  - Rochester, New York
  - Charlotte, North Carolina
  - Winston-Salem, North Carolina
  - Penndel, Pennsylvania
  - Johnston, Rhode Island
  - Mt. Pleasant, South Carolina
  - Simpsonville, South Carolina
  - Colleyville, Texas
  - Houston, Texas
  - San Antonio, Texas

REFERENCES:
- [Result] Thakkar RB, Kashyap ML, Lewin AJ, Krause SL, Jiang P, Padley RJ. Acetylsalicylic acid reduces niacin extended-release-induced flushing in patients with dyslipidemia. Am J Cardiovasc Drugs. 2009;9(2):69-79. doi: 10.1007/BF03256578. PMID 19331435

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 47 study sites in the United States between February and April, 2008.
Pre-assignment Details: This study had a 1-week run-in (acetylsalicylic acid [ASA] 325 mg or ASA placebo [Pbo] once daily) prior to 4 weeks of niacin extended-release (NER) plus ASA/ASA Pbo coadministration. Ten of 277 randomized subjects discontinued before run-in due to withdrawal of consent (4), lost to follow-up (4), protocol violation (1), and other (1).
Groups:
- NER 500; ASA run-in, ASA Coadmin: Aspirin (ASA) 325 mg daily during run-in (1 week); ASA 325 mg 30 min prior to niacin extended-release ([NER], 500 mg starting dose), daily during coadministration (4 weeks)
- NER 500; ASA Pbo run-in, ASA Coadmin: Aspirin placebo (ASA Pbo) daily during run-in (1 week); ASA 325 mg 30 min prior to niacin extended-release ([NER], 500 mg starting dose), daily during coadministration (4 weeks)
- NER 500; ASA Pbo run-in, ASA Pbo Coadmin: Aspirin placebo (ASA Pbo) daily during run-in (1 week); ASA Pbo 30 min prior to niacin extended-release ([NER], 500 mg starting dose), daily during coadministration (4 weeks)
- NER 1000; ASA run-in; ASA Coadmin: Aspirin (ASA) 325 mg daily during run-in (1 week); ASA 325 mg 30 min prior to niacin extended-release ([NER], 1000 mg starting dose), daily during coadministration (4 weeks)
- NER 1000; ASA Pbo run-in, ASA Coadmin: Aspirin placebo (ASA Pbo) daily during run-in (1 week); ASA 325 mg 30 min prior to niacin extended-release ([NER], 1000 mg starting dose), daily during coadministration (4 weeks)
- NER 1000; ASA Pbo run-in, ASA Pbo Coadmin: Aspirin placebo (ASA Pbo) daily during run-in (1 week); ASA Pbo 30 min prior to niacin extended-release ([NER], 1000 mg starting dose), daily during coadministration (4 weeks)
Period: Run-in Period
Arm/Group | NER 500; ASA run-in, ASA Coadmin | NER 500; ASA Pbo run-in, ASA Coadmin | NER 500; ASA Pbo run-in, ASA Pbo Coadmin | NER 1000; ASA run-in; ASA Coadmin | NER 1000; ASA Pbo run-in, ASA Coadmin | NER 1000; ASA Pbo run-in, ASA Pbo Coadmin
Started | 45 | 44 | 44 | 44 | 45 | 45
Completed | 44 | 43 | 41 | 43 | 41 | 44
Not Completed | 1 | 1 | 3 | 1 | 4 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 1 | 3 | 1
Not completed — Noncompliance | 1 | 0 | 1 | 0 | 0 | 0
Period: Coadministration Period
Arm/Group | NER 500; ASA run-in, ASA Coadmin | NER 500; ASA Pbo run-in, ASA Coadmin | NER 500; ASA Pbo run-in, ASA Pbo Coadmin | NER 1000; ASA run-in; ASA Coadmin | NER 1000; ASA Pbo run-in, ASA Coadmin | NER 1000; ASA Pbo run-in, ASA Pbo Coadmin
Started | 44 | 43 | 41 | 43 | 41 | 44
Completed | 40 | 38 | 31 | 36 | 36 | 38
Not Completed | 4 | 5 | 10 | 7 | 5 | 6
Not completed — Adverse Event | 3 | 1 | 7 | 4 | 3 | 4
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 1 | 0 | 1
Not completed — Protocol Violation | 0 | 1 | 0 | 1 | 1 | 0
Not completed — Other | 0 | 2 | 3 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- NER 1000; ASA run-in, ASA Coadmin: Aspirin (ASA) 325 mg daily during run-in (1 week); ASA 325 mg 30 min prior to niacin extended-release ([NER], 1000 mg starting dose), daily during coadministration (4 weeks)
- Total: Total of all reporting groups
Arm/Group | NER 500; ASA run-in, ASA Coadmin | NER 500; ASA Pbo run-in, ASA Coadmin | NER 500; ASA Pbo run-in, ASA Pbo Coadmin | NER 1000; ASA run-in, ASA Coadmin | NER 1000; ASA Pbo run-in, ASA Coadmin | NER 1000; ASA Pbo run-in, ASA Pbo Coadmin | Total
Number analyzed (Participants) | 44 | 43 | 41 | 43 | 41 | 44 | 256
Age Continuous [Mean (Standard Deviation); unit: Years] — Includes only those subjects who entered the coadministration period and received at least one dose of study medication.
  Years | 55.5 (10.62) | 49.0 (10.48) | 51.5 (12.58) | 53.7 (12.4) | 54.8 (11.08) | 52.3 (12.45) | 52.8 (11.73)
Sex: Female, Male [Count of Participants; unit: Participants] — Includes only those subjects who entered the coadministration period and received at least one dose of study medication.
  Participants
    Female | 21 | 23 | 21 | 15 | 21 | 23 | 124.0
    Male | 23 | 20 | 20 | 28 | 20 | 21 | 132.0
Region of Enrollment [Number; unit: participants] — Includes only those subjects who entered the coadministration period and received at least one dose of study medication.
  participants
    United States | 44 | 43 | 41 | 43 | 41 | 44 | 256.0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Severity of Flushing Events During Week 1 of Niacin Extended-release (NER) Treatment
Description: The maximum severity of flushing events subjects experienced during Week 1 of NER treatment was categorized as none, mild, moderate, severe, or very severe using the Flushing Assessment Tool via an e-diary. Flushing was assessed daily and the percentage of subjects with maximum flushing severity in each category was calculated.
Time Frame: From Baseline to end of Week 1
Population: All subjects in the modified intent-to-treat population, defined as all subjects who took at least 1 dose of study medication and who had at least 1 entry in the Flushing Assessment Tool e-diary (n = 251).
Measure: Number; unit: Percentage of Subjects
Groups:
- Any Acetylsalicylic Acid: Pooled arms that received acetylsalicylic acid (ASA) 325 mg during run-in and/or coadministration.
- No Acetylsalicylic Acid: Pooled arms that received acetylsalicylic acid placebo (ASA Pbo) during run-in and coadministration.
Arm/Group | Any Acetylsalicylic Acid | No Acetylsalicylic Acid
Number analyzed (Participants) | 167 | 84
Percentage of Subjects
  None | 57 | 48
  Mild | 28 | 24
  None/mild | 85 | 71
  Moderate | 11 | 17
  Severe | 4 | 8
  Very severe | 1 | 4
Statistical Analysis 1: Comparison: Any Acetylsalicylic Acid vs No Acetylsalicylic Acid; Test type: Superiority or Other; p = 0.010, Cochran-Mantel-Haenszel — No adjustments were made for multiple comparisons. P-values <= 0.05 were reported as statistically significant

2. Secondary Outcome: Maximum Severity of Flushing Events Overall During 4 Weeks of Niacin Extended-release (NER) Treatment
Description: The maximum severity of flushing events subjects experienced during 4 weeks of NER treatment was categorized as none, mild, moderate, severe, or very severe using the Flushing Assessment Tool via an e-diary. Flushing was assessed daily and the percentage of subjects with maximum flushing severity in each category was calculated.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of Subjects
Arm/Group | Any Acetylsalicylic Acid | No Acetylsalicylic Acid
Number analyzed (Participants) | 167 | 84
Percentage of Subjects
  None | 30 | 15
  Mild | 28 | 14
  None/Mild | 58 | 30
  Moderate | 28 | 35
  Severe | 11 | 23
  Very severe | 4 | 13

3. Secondary Outcome: Mean of Maximum Severity of Flushing Events Overall During 4 Weeks of Niacin Extended-release (NER) Treatment
Description: Subjects assessed the severity of flushing events on a 10-point numeric rating scale of 1-3 (mild), 4-6 (moderate), 7-9 (severe), and 10 (very severe) using the Flushing Assessment Tool via an e-diary. For subjects who did not experience flushing, a score of 0 was assigned. Flushing was assessed daily.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Any Acetylsalicylic Acid | No Acetylsalicylic Acid
Number analyzed (Participants) | 167 | 84
Scores on a Scale | 3.1 (2.86) | 5.1 (3.16)

4. Secondary Outcome: Mean Number of Moderate or Greater Flushing Events Per Subject Per Week Overall During 4 Weeks of Niacin Extended-release (NER) Treatment
Description: Flushing was assessed daily using the Flushing Assessment Tool via an e-diary and the mean number of flushing events per subject per week considered moderate or greater in severity was calculated. Flushing events were rated by the subject using a categorical scale of mild, moderate, severe, or very severe.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of Events per Subject per Week
Arm/Group | Any Acetylsalicylic Acid | No Acetylsalicylic Acid
Number analyzed (Participants) | 167 | 84
Number of Events per Subject per Week | 0.3 (0.64) | 0.8 (1.10)

ADVERSE EVENTS:
Arm/Group | Any Acetylsalicylic Acid | No Acetylsalicylic Acid
Serious Adverse Events (participants affected / at risk) | 1 | 1
Other Adverse Events (participants affected / at risk) | 119 | 72
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Any Acetylsalicylic Acid | No Acetylsalicylic Acid
Esophageal ulcer (Gastrointestinal disorders) | 0/171 (0) | 1/85 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1/171 (1) | 0/85 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Any Acetylsalicylic Acid | No Acetylsalicylic Acid
Nausea (Gastrointestinal disorders) | 4/171 | 1/85
Non-cardiac chest pain (General disorders) | 1/171 | 2/85
Blood creatine phosphokinase increased (Investigations) | 0/171 | 2/85
Blood uric acid increased (Investigations) | 0/171 | 2/85
Arthralgia (Musculoskeletal and connective tissue disorders) | 1/171 | 3/85
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0/171 | 2/85
Rash (Skin and subcutaneous tissue disorders) | 3/171 | 2/85
Flushing (Vascular disorders) | 117/171 | 71/85

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Provide Abbott at least sixty (60) days prior to submission for review, Abbott shall return comments within sixty (60) days of receipt of draft. Proposed draft shall be delayed an additional sixty (60) days in addition to the Review Period.